CLINICAL TRIAL: NCT06408636
Title: Cardiac MRI Left Atrial Strain Associated With Ischemic Stroke in Patients With Acute Myocardial Infarction
Brief Title: Prognostic Role of LA Strain in Acute Myocardial Infarction
Acronym: CMR-MI
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2023-KL222-01
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Myocardial Infarction, Acute; Stroke Ischemic; Mortality
Keywords: cardiac magnetic resonance; myocardial infarction; atrial fibrillation; ischemic stroke
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Infarction; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- We consecutively selected patients diagnosed with acute myocardial infarction from September 2019 th
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI — All selected patients completed a cardiac magnetic resonance examination without other interventions.

SUMMARY:
This is a single-center retrospective observational study in which we consecutively selected patients diagnosed with acute myocardial infarction from September 2019 to March 2024 at the Affiliated Hospital of Xuzhou Medical University. Inclusion criteria: 1. CMR was completed during all hospitalizations; 2. complete clinical data; 3. received continuous cardiac monitoring during hospitalization. Exclusion criteria: 1. unclear or non-compliant CMR images; 2. previous history of myocardial infarction; 3. malignant tumors diseases. Dedicated cardiovascular imaging software CVI42 (cvi42® version 5.13.5, Circle Cardiovascular Imaging, Canada) was used for image analysis. LA strain was obtained by cardiac MRI feature tracking. Patient prognosis was obtained through chart notes and telephone follow-up. Major events included atrial fibrillation, ischemic stroke, and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* 1.CMR was completed during all hospitalizations; 2. complete clinical data; 3. received continuous cardiac monitoring during hospitalization.

Exclusion Criteria:

* 1.unclear or non-compliant CMR images; 2. previous history of myocardial infarction; 3. malignant tumors diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a single-center retrospective observational study in which we consecutively selected patients diagnosed with acute myocardial infarction from September 2019 to March 2024 at the Affiliated Hospital of Xuzhou Medical University. Dedicated cardiovascular imaging software CVI42 (cvi42® version 5.13.5, Circle Cardiovascular Imaging, Canada) was used for image analysis. LA strain was obtained by cardiac MRI feature tracking. Patient prognosis was obtained through chart notes and telephone follow-up. Major events included atrial fibrillation, ischemic stroke, and all-cause mortality.
Sampling Method: Probability Sample
Enrollment: 780 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint events included all-cause death, ischemic stroke, and atrial fibrillation | All patients were followed until March 31, 2024

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No